CLINICAL TRIAL: NCT02889744
Title: Comparison of Cerebral Tissue Oxygen Saturation (SctO2) Between 36℃ and 33℃ of Targeted Temperature Management (TTM) After Cardiac Arrest
Brief Title: Comparison of Cerebral SctO2 Between 36℃ and 33℃ of TTM After Cardiac Arrest
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: Bard Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: SNUH0620160330
Record Dates: First submitted 2016-08-18; First posted 2016-09-07 (Estimated); Last update posted 2021-03-18 (Actual); Status verified 2021-03

CONDITIONS: Heart Arrest
Keywords: Temperature; Hypothermia; Brain; Oxygen; Prognosis
MeSH Terms: conditions — Heart Arrest; Hypothermia

STUDY DESIGN:
Intervention Model Description: From the results of previous studies, we assumed that the mean difference in rSO2 at 72 h between the 36℃ or 33℃ groups would be 3% with 4% of standard deviation. By a referral (2015-0207) to the Medical Research Collaborating Center (MRCC) of SNUH/SNUMC, a sample size of at least 58 (29 per group) was calculated with a power of 0.8 and a significance level of 0.05. Considering an unexpected loss of 15%, the study was planned for 66 participants.
  Randomization was performed by the 4, 6-block randomization method at the MRCC SNUH/SNUMC web-site (http://mrcc.snu.ac.kr).
Who Masked: Outcomes Assessor
Masking Description: Primary and secondary outcomes were assessed by an investigator blinded to this study.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 36-TH (Active Comparator): Core temperature 36℃ of targeted temperature management (36-TH) for 24 hours in cardiac arrest victims using Arctic Sun.
  Interventions: Device: Arctic Sun
- 33-TH (Active Comparator): Core temperature 33℃ of targeted temperature management (36-TH) for 24 hours in cardiac arrest victims using Arctic Sun.
  Interventions: Device: Arctic Sun

INTERVENTIONS:
Device: Arctic Sun — Targeted temperature management for 24 hours with core temperature 36℃ or 33℃
  Other Names: External cooling device

SUMMARY:
The investigators hypothesize that

1. if decrease in SctO2 level is caused by the degree of hypothermia, SctO2 level in the 33-TH may be lower than that in the 36-TH group.
2. if decrease in SctO2 level is not caused by the degree of hypothermia but caused by brain injury, SctO2 level may be associated with only the prognosis of cardiac arrest victims regardless of core temperatures.

The primary objective of this study is to compare the 72-hour changes in SctO2 level between the 36-TH and 33-TH groups in cardiac arrest victims.

DETAILED DESCRIPTION:
1. Subject Identification and Screening For each cohort, patients will be identified after acquisition of sustained return of spontaneous circulation (ROSC) (> 30 minutes). If the patients meet inclusion/exclusion criteria, patients will be enrolled in the study. The investigators will obtain written informed consent from all of the patients or their representatives.
2. Assignment of Subject Number A unique identification number will be given to study subjects in an attempt to de-identify their information. Subject numbers will be assigned in sequential order. The subject number will consist of four digits. The first two digits will designate the study site. The last two digits will designate the subject by number in sequential order (i.e., subject number 01 01 will be the first subject at site 1; 01 02 will be the second subject at site 1, etc.).
3. Study Methods

   * Randomization to 36-TH (core body temperature (BT) 36℃) or 33-TH (core BT 33℃) group will be performed by a web based randomization site (http://mrcc.snuh.org).
   * Start target temperature management using external cooling device (Arctic Sun) within 1 hour post-ROSC.
   * SctO2 monitoring starts within 1 hour post-ROSC and maintain for 72 hours.
   * 36-TH (core BT 36℃) or 33-TH (core BT 33℃) for 24 hours
   * Rewarming 0.25℃/h in 33-TH group
   * Core temperature < 37.5℃ for 72 hours

   All patients will be treated per the postresuscitation care protocol. Target treatment will include
   * Target: central venous pressure (CVP) (8 - 12 mmHg), mean arterial pressure (MAP) (> 65 mmHg), central venous oxygen saturation (ScvO2) (> 70%)
   * Seizure control, shivering control as appropriate
   * Coronary intervention as soon as possible if needed
   * Infection control if indicated
   * Other supportive care

   Monitoring data including
   * CVP, MAP, ScvO2, lactate, neuron specific enolase (NSE), end-tidal carbon dioxide (EtCO2), input-output (I/O) balance
   * Intermittent electroencephalography (EEG) monitoring (2 times/72 hours)
   * Laboratory data including arterial blood gas analysis (ABGA), complete blood count (CBC), liver function test (LFT), electrolyte, blood urea nitrogen/creatinine (BUN/Cr), et al.
   * SctO2
   * Core (esophageal or bladder) temperature
4. Data Collection

Study data will be collected in the following manner:

• All data will be collected on appropriate Case Report Forms.

ELIGIBILITY:
Inclusion Criteria:

* Comatose patients successfully resuscitated from cardiac arrest

Exclusion Criteria:

* < 18 years old
* Definite non-cardiac cause arrest
* Contraindication to TH Active bleeding, coagulopathy, fatal arrhythmia, severe infectious condition
* Presence of advanced directives to withhold or withdraw life-sustaining treatment
* Expected survival < 72 hours
* Underlying low CPC (≤ 3)
* No informed consent
* Follow-up loss

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2016-03; Primary Completion 2020-07 (Actual); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
The comparison of the 72-hour SctO2 level between the 36-TH and 33-TH groups in cardiac arrest victims | 72 hour

SECONDARY OUTCOMES:
The comparison of the 72-hour changes in SctO2 level between the 36-TH and 33-TH groups | 0, 24, and 72 hours
The comparison of the severity scores between the 36-TH and 33-TH groups | 0, 24, and 72 hours
  * APACHE II score
  * Sequential Organ Failure Assessment (SOFA) score
The comparison of the serum biomarker levels between the 36-TH and 33-TH groups | 0, 24, and 72 hours
  * Neuron specific enolase
  * Cytokines
  * Antioxidants
The comparison of the number of patients with survival discharge between the 36-TH and 33-TH groups | 6 months
The comparison of the 6-month cerebral performance scale (CPC) between the 36-TH and 33-TH groups | 6 months
Complication of therapeutic hypothermia | 72 hours
  * Bleeding requiring transfusion
  * Fatal arrhythmia requiring intervention
  * Electrolyte imbalance: newly developed abnormal values
  * Hyper/hypoglycemia
  * Sepsis/pneumonia

CONTACTS AND LOCATIONS:
Overall Officials: Gil Joon Suh, MD, PhD, Principal Investigator — Seoul National Univerisity College of Medicine
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hypothermia after Cardiac Arrest Study Group. Mild therapeutic hypothermia to improve the neurologic outcome after cardiac arrest. N Engl J Med. 2002 Feb 21;346(8):549-56. doi: 10.1056/NEJMoa012689. PMID 11856793
- [Background] Nielsen N, Wetterslev J, Cronberg T, Erlinge D, Gasche Y, Hassager C, Horn J, Hovdenes J, Kjaergaard J, Kuiper M, Pellis T, Stammet P, Wanscher M, Wise MP, Aneman A, Al-Subaie N, Boesgaard S, Bro-Jeppesen J, Brunetti I, Bugge JF, Hingston CD, Juffermans NP, Koopmans M, Kober L, Langorgen J, Lilja G, Moller JE, Rundgren M, Rylander C, Smid O, Werer C, Winkel P, Friberg H; TTM Trial Investigators. Targeted temperature management at 33 degrees C versus 36 degrees C after cardiac arrest. N Engl J Med. 2013 Dec 5;369(23):2197-206. doi: 10.1056/NEJMoa1310519. Epub 2013 Nov 17. PMID 24237006
- [Result] Buunk G, van der Hoeven JG, Meinders AE. A comparison of near-infrared spectroscopy and jugular bulb oximetry in comatose patients resuscitated from a cardiac arrest. Anaesthesia. 1998 Jan;53(1):13-9. doi: 10.1111/j.1365-2044.1998.00263.x. PMID 9505736
- [Result] Suffoletto B, Kristan J, Rittenberger JC, Guyette F, Hostler D, Callaway C. Near-infrared spectroscopy in post-cardiac arrest patients undergoing therapeutic hypothermia. Resuscitation. 2012 Aug;83(8):986-90. doi: 10.1016/j.resuscitation.2012.03.021. Epub 2012 Apr 19. PMID 22521725
- [Result] Meex I, Dens J, Jans F, Boer W, Vanhengel K, Vundelinckx G, Heylen R, De Deyne C. Cerebral tissue oxygen saturation during therapeutic hypothermia in post-cardiac arrest patients. Resuscitation. 2013 Jun;84(6):788-93. doi: 10.1016/j.resuscitation.2013.01.003. Epub 2013 Jan 8. PMID 23313422